CLINICAL TRIAL: NCT03242447
Title: Evaluation of e-Practice Self-Regulation (e-PS-R)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Policy & Research Group (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 90AP2679-01-00
Record Dates: First submitted 2017-07-25; First posted 2017-08-08 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Teen Pregnancy Prevention

STUDY DESIGN:
Intervention Model Description: participants are assigned to one of two or more groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-Practice Self-Regulation (e-PS-R) (Experimental): e-Practice Self-Regulation (e-PSR) is the treatment condition. e-PS-R is a 'blended learning' intervention, combining online and face-to-face instruction. e-PS-R aims to increase knowledge of sexual health and the impact of trauma on sexual decision-making.
  Interventions: Behavioral: e-Practice Self-Regulation
- Video Health Group (Active Comparator): The Video Health Group is the control counterfactual condition. Youth assigned to the control group will view a video on a non-sexual health topic (the hazards of smoking).The video for the control condition will be The Toxic Life Cycle of a Cigarette, a 17-minute video that details the negative effects that cigarettes have on the environment and on people who manufacture and use cigarettes. The informational video uses both narration and interviews to educate viewers on the dangers that cigarettes pose.
  Interventions: Behavioral: Video Health Group

INTERVENTIONS:
Behavioral: e-Practice Self-Regulation — e-PS-R utilizes 'blended learning', the combination of online and face-to-face instruction, and incorporates online videos and interactive elements that have been shown to be effective with high-risk youth. e-PS-R consists of eight 30-minute e-learning sessions for youth participants and four 30-45 minute one-on-one in-person meetings between youth and a trained facilitator.
  Arms: e-Practice Self-Regulation (e-PS-R)
Behavioral: Video Health Group — The video for the control condition will be The Toxic Life Cycle of a Cigarette, a 17-minute video that details the negative effects that cigarettes have on the environment and on people who manufacture and use cigarettes.
  Arms: Video Health Group

SUMMARY:
The purpose of the study is to determine the impact of the offer to participate in the e-Practice Self-Regulation (e-PS-R) (treatment) relative to the control condition on increasing knowledge of sexual health and the impact of trauma on sexual decision-making and preventing teen pregnancy and high-risk behaviors 12 months after enrollment.

DETAILED DESCRIPTION:
The Policy & Research Group (PRG) will be conducting a rigorous evaluation of an innovative intervention designed to prevent adolescent pregnancy, births, and STIs among high-risk youth populations, entitled online Practice Self-Regulation (e-PS-R). e-PS-R is the online adaptation of the Practice Self-Regulation (PS-R); both PS-R and e-PS-R were developed through grant funding by Joann Schladale of Resources for Resolving Violence, Inc. The original PS-R intervention is a 10-session therapeutic program designed for youth ages 14-19 who have experienced trauma; each session is intended to be offered by a masters-level therapist during one-on-one weekly therapy sessions. The online adaptation e-PS-R utilizes 'blended learning', the combination of online and face-to-face instruction, and incorporates online videos and interactive elements that have been shown to be effective with high-risk youth. e-PS-R consists of eight 30-minute e-learning sessions for youth participants and four 30-45 minute one-on-one in-person meetings between youth and a trained facilitator. The following Adulthood Preparation Subjects are covered during both the online sessions and the in-person meetings: Adolescent Development, Healthy Life Skills, and Healthy Relationships. By increasing knowledge of sexual health and the impact of trauma on sexual decision-making, the program is designed to encourage and support youth in practicing self-regulation.

The Policy & Research Group (PRG) will conduct an implementation evaluation and an impact evaluation, using a randomized controlled trial, to test the effectiveness of this new intervention. The study will target juvenile justice-involved youth ages 14-19 who have experienced trauma. The primary focus of the study will be to investigate the impact of the intervention on two self-reported sexual behaviors: (1) inconsistency of condom use, and (2) number of sexual partners. In addition, the study will include exploratory investigations of the following self-reported sexual behaviors and theoretically relevant antecedents to behavior and pathways to behavior change: (1) use of contraception; (2) use of dual methods of protection; (3) incidence of pregnancy; (4) self-efficacy to engage in affect regulation; (5) sexual self-efficacy; (6) intentions to engage in affect-regulation; (7) intentions to engage in sexual self-regulation; and (8) use of affect regulation. Outcomes will be assessed using self-reported, participant-level data gathered (by way of a questionnaire) at four time points: baseline (enrollment); post-program (immediately after the end of the intervention period; 3 months after baseline); short-term (3 months post-intervention period) follow-up; and long-term (nine months post-intervention period) follow-up.

Starting in July 2017 and continuing for two years, 600 participants will be enrolled into the study at partner implementation sites within the juvenile justice systems in New Mexico and West Virginia. The third and fourth years of the grant will be used to complete the following tasks: collect follow-up data from study participants; conduct implementation and impact evaluation analysis, reporting, and dissemination efforts; and manualize and package the curriculum and training materials.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 14-19
* Be involved with the juvenile justice system
* Be deemed appropriate for study by site staff and study facilitator (no acute illness or behavioral problems; psychiatrically stable; cognitively capable of internalizing and comprehending content of intervention)
* Possess adequate English-language comprehension (be able to read and comprehend the on-line intervention materials, which are available only in English)
* Consent/assent to participating in study

Exclusion Criteria:

* Not be residing in or scheduled to enter a secure facility
* Not be currently pregnant
* Not be trying to get pregnant
* Not be an enrolled participant (former or current) in the Teen Health Study (Teen Pregnancy Prevention study funded by the Office of Adolescent Health, being conducted in Albuquerque, New Mexico)
* Not have previously participated in e-PS-R

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 631 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
participants' self-reported sexual behaviors | 12 months after enrollment into the study
  The primary outcome will be the mean differences between the treatment and control group participants in self-reported sexual behaviors at 12-month follow-up; exploratory analyses will examine differences in sexual behaviors post-program and differences in other theoretically relevant outcomes (e.g., attitudes, self-efficacies, self-regulatory behaviors) at both post-program and 12-month follow-up.
  The independent variable of interest will be the treatment assignment, which will be operationalized as being randomly assigned to the active treatment (1) or the control condition (0).

SECONDARY OUTCOMES:
consistency of contraceptive use | 12 months after enrollment
  The risk outcome is operationalized as the proportion of times a person reports having sexual intercourse without using any form of birth control (including condoms). The measure is calculated from the following items:
  The measure is calculated by dividing the total number of times a person reported having sexual intercourse without using any contraception by the total number of times she reported having sexual intercourse.
  The resulting variable is a continuous proportion with values that range from 0 to 1, where 0 indicates that a person has not engaged in sexual intercourse without birth control in the past three months, and 1 indicates that the person has engaged in sexual intercourse without birth control (risk behavior) 100% of the times they had sex in the past three months.
frequency of sexual activity | 12 months after enrollment
  The risk outcome is operationalized as the number of times in the past three months a person reports having any type of sex.
  The measure is taken directly from the following item:
  • In total, how many times have you had any type of sex in the past 3 months?
  The variable is continuous, with values ranging from 0 to k, where 0= no sexual activity reported in past 3 months and k = number of times sex reported.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jenner, PhD, Principal Investigator — The Policy & Research Group
Locations (1):
- The Policy & Research Group, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A dataset will be prepared at the conclusion of the study, which includes de-identified individual-level data on all study participants who contributed self-report data. Respondents will be represented only by a research ID number. Included in the dataset will be self-report data collected across all survey administrations (including demographic characteristics, sexual behaviors, and theoretical antecedents to those behaviors) and select information on program participation (e.g., which program sessions were attended). Basic data cleaning steps will be taken in order to ensure data are unidentifiable and to increase usability.
Time Frame: The individual participant dataset will become available twelve months after the study has concluded.